CLINICAL TRIAL: NCT00622739
Title: Ziprasidone in Pediatric Bipolar Disorder: a 6-week, Open-label Comparison of Rapid vs. Slow Dose Titration
Brief Title: Ziprasidone in Pediatric Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Stanley Medical Research Institute (Other); Pfizer (Industry); Children's Medical Center Dallas (Other)
Responsible Party: Principal Investigator, Kirti Saxena, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaxenaZiprasidone
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Children; Adolescents; Treatment
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ziprasidone rapid dose (Active Comparator): Rapid Dose Titration Group
  Interventions: Drug: Ziprasidone
- ziprasidone slow dose (Active Comparator): Slow Dose Titration Group
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Subjects will be treated openly with Ziprasidone for 6 weeks. Dose will be titrated from 20 mg to a maximum of 160 mg. Arm 1 will have the dose of Ziprasidone titrated at a rate of 20 mg every 2 days, reaching the maximum dose in 14 days. Final dose of Ziprasidone will be determined by symptoms reduction and the presence or absence of side effects.
  Other Names: Geodon
  Arms: ziprasidone rapid dose
Drug: Ziprasidone — Subjects will be treated openly with Ziprasidone for 6 weeks. Dose will be titrated from 20mg to a maximum of 160mg. Arm 2 will have the dose of Ziprasidone titrated at a rate of 20mg every 3-4 days, reaching the maximum dose in 25 days. Final dose of Ziprasidone will be determined by symptoms reduction and the presence or absence of side effects.
  Other Names: Geodon
  Arms: ziprasidone slow dose

SUMMARY:
This is a 6 week, open-label, blinded-rater, randomized, controlled, pilot study designed to determine the dosing, safety and efficacy of ziprasidone in the treatment of pediatric bipolar disorder (PBD). In this pilot study we are comparing the efficacy of rapid versus slow dose titration of ziprasidone in PBD. The investigators hypothesize that subjects on ziprasidone monotherapy will have a reduction in manic symptoms. Also, the investigators hypothesize that slower titration of ziprasidone will result in lesser side effects which will assist in medication compliance as measured by patient report and pill count.

DETAILED DESCRIPTION:
This study will enroll approximately 60 children and adolescents aged 10-17 years who have been diagnosed with bipolar disorder. Their participation will last about 8 weeks (2 weeks of screening and 6 weeks of medication management) and enrollment will last for two years. After the screening period, all subjects who meet inclusion/exclusion criteria will be randomized to either rapid or slow dose titration of ziprasidone. Subjects in the rapid titration group will reach their maximum dose of study drug over 2 weeks, subjects in the slow titration group over 4 weeks. The study doctor may deviate from the dosing schedule if clinically indicated. The primary data analysis of this pilot study will examine the effect of rapid- versus slow-dose titration of ziprasidone on manic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 10-17 years
* Currently meet Diagnostic and Statistical Manual of Mental Disorders IV-Text Revision (DSM-IV-TR) criteria for bipolar disorder, type I, II or Not Otherwise Specified (NOS) as determined by the Schedule for Affective Disorders and Schizophrenia -Present/Lifetime (Kiddie-SADS-PL)
* Experiencing manic, hypomanic or mixed states as determined by clinical diagnosis and Kiddie- Young Mania rating scale (K-YMRS) equal to or more than 14
* General good health as determined by medical history, physical examination, and laboratory evaluations
* Female adolescents, if sexually active, must practice birth control methods approved by the primary investigator
* Ability to swallow tablets
* Subject's parent or guardian must be fully capable of monitoring the subject's disease process and compliance to treatment
* Parent(s) or legal guardian(s) must read and sign the informed consent form after the nature of the study has been fully explained and assent must be obtained from subjects.

Exclusion Criteria:

* Have a lifetime DSM-IV-TR Axis I disorder diagnosis of autistic disorder, schizophrenia, schizoaffective disorder, or other psychotic disorders
* DSM-IV-TR diagnosis of alcohol or substance abuse or dependence within the past 6 months
* Serious or unstable medical or neurological conditions which require concomitant medications
* Judged by the principal investigator (PI) to be acutely suicidal or homicidal, or at imminent risk of injuring self or others or causing significant damage to property-i.e., subject needs to be in an inpatient facility
* Known or suspected intelligence quotient (IQ) less than 70
* Have a DSM-IV-TR diagnosis of anorexia and/or bulimia at the time of screening or within the last six months
* Female who is pregnant or nursing
* Subjects with a history of syncopal episodes (sudden loss of consciousness with loss of postural tone and not preceded by a pre-syncopal phase) or unexplained loss of consciousness
* Subjects with a history of significant cardiovascular disease or significant concurrent cardiovascular disease, including uncontrolled hypertension, hypotension, congestive heart failure or congenital heart disease
* Subjects with a history of cardiac arrhythmias, conduction abnormalities or known personal history or corrected QT prolongation (including congenital long QT syndrome)
* Subjects with a known genetic risk for QT syndrome determined by family history in first degree relatives
* Subjects taking any medications known to interact with ziprasidone or subjects taking any medications which have been consistently observed to prolong the QT interval
* Subjects with a clinically significant ECG abnormality at screening
* Subjects with persistent QTc (Fridericia) * 460 msec at screening
* Screening laboratory values outside the normal range and judged to be clinically significant by the investigator
* Patients and families that are Spanish speaking only will be excluded from the study as some instruments used in the study have not been validated in Spanish

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Saxena, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone Rapid Dose Group: Rapid Dose Titration Group
  Ziprasidone: Subjects will be treated openly with Ziprasidone for 6 weeks. Dose will be titrated from 20 mg to a maximum of 160 mg. Arm 1 will have the dose of Ziprasidone titrated at a rate of 20 mg every 2 days, reaching the maximum dose in 14 days. Final dose of Ziprasidone will be determined by symptoms reduction and the presence or absence of side effects.
- Ziprasidone Slow Dose Group: Slow Dose Titration Group
  Ziprasidone: Subjects will be treated openly with Ziprasidone for 6 weeks. Dose will be titrated from 20mg to a maximum of 160mg. Arm 2 will have the dose of Ziprasidone titrated at a rate of 20mg every 3-4 days, reaching the maximum dose in 25 days. Final dose of Ziprasidone will be determined by symptoms reduction and the presence or absence of side effects.
Period: Overall Study
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Started | 13 | 15
Completed | 11 | 9
Not Completed | 2 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 13.53 (2.62) | 13.38 (2.50) | 13.4 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) is a measure of the severity of manic symptoms. The scores on the scale range from 0-56. A score of more than or equal to 14 was the cut off for inclusion into this study. A higher score denotes increased severity of manic symptoms.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Number analyzed (Participants) | 13 | 15
units on a scale | 12.70 (1.41) | 12.57 (1.32)

2. Secondary Outcome: Children's Depression Rating Scale
Description: The CDRS-R is a 17 item clinician-rated instrument used to measure severity of depressive symptoms in youth (ages 6-18). Each item is rated on a 1 to 5 or 1 to 7 point scale, with a 1 describing absence of the given symptom. The CDRS-R yields a total score from 17 to 113 with a score of 40 or greater considered to symptomatic of depression. Scores of 35-40 indicate mild depression, 29-34 is borderline and <28 is no depression.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ziprasidone Rapid Dose | Ziprasidone Slow Dose
Number analyzed (Participants) | 13 | 15
score on a scale | 32.56 (1.44) | 29.22 (1.34)

3. Secondary Outcome: Clinical Global Impressions-Severity (CGI-S) Scale
Description: The CGI-S assesses clinical severity. The CGI-S is a seven point scale where 1 is the minimum value and 7 is the maximum value. Lower scores mean a better outcome.
  The CGI-Severity scale scores are: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone Rapid Dose | Ziprasidone Slow Dose
Number analyzed (Participants) | 13 | 15
units on a scale | 3.63 (0.19) | 3.36 (0.18)

4. Secondary Outcome: SAFTEE (Side Effects Rating Scale)
Description: The Systematic Assessment for Treatment of Emergent Events (SAFTEE) is one of the first comprehensive Adverse effects-elicitation instruments developed specifically for use in psychiatric clinical trials. The SAFTEE is a standardized method, which increases consistency of Adverse Effects data, both within and across clinical trials.It allows ratings of five levels of severity and collects information about the onset, duration, pattern, judgement of attribution of cause, and action taken by the clinician. Suggested probe questions are also provided, which the clinician can use to elicit detailed information about the AE. Furthermore, the SAFTEE requires the clinician to determine a time interval of inquiry to be used in the trial. Adverse Effects are graded as None=0, Mild=1, Moderate=2, Severe=3.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Number analyzed (Participants) | 13 | 15
units on a scale | 0.32 (0.09) | 0.46 (0.08)

5. Secondary Outcome: AIMS (Abnormal Involuntary Movement Scale)
Description: AIMS is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs, such as tardive dystonia and chronic akathisia, as well as 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in three main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe).
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Number analyzed (Participants) | 13 | 15
units on a scale | 0.20 (0.15) | 0.32 (0.14)

6. Secondary Outcome: Barnes Akathisia Rating Scale (BARS)
Description: The BARS measures drug-induced akathisia occurring specifically with use of neuroleptic agents. It is a four-item fully anchored scale. Three items (objective akathisia, subjective awareness of restlessness, and subjective distress related to restlessness) are rated on a 4-point scale (0= normal and 9= most severe) and, the global clinical assessment of akathisia uses a 5-point scale (0= normal and 4= most severe).
  Total scores ranged from 0-13 with higher scores reflecting more akathisia.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Number analyzed (Participants) | 13 | 15
units on a scale | 0.11 (0.05) | 0.06 (0.04)

ADVERSE EVENTS:
Arm/Group | Ziprasidone Rapid Dose Group | Ziprasidone Slow Dose Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 1/13 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone Rapid Dose Group (N=13) | Ziprasidone Slow Dose Group (N=15)
Dystonic Reaction (Psychiatric disorders) | 1 (1) | 0 (0)
worsening of mood and inadequate response to medicaiton (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No